CLINICAL TRIAL: NCT04011462
Title: Perioperative Normothermia: Temperature and Prewarming Methods
Acronym: Normothermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Vanessa de Brito Poveda, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VPoveda
Record Dates: First submitted 2019-05-21; First posted 2019-07-08 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Hypothermia
Keywords: Nursing; Hypothermia; Perioperative Nursing
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prewarming 20 minutes (Experimental): prewarming with a forced air warming system, using a blanket covering the whole body, regulated to the temperature of 38 °C for 20 minutes.
  Interventions: Device: prewarming 20 minutes
- Prewarming 30 minutes (Experimental): prewarming with a forced air warming system, using a blanket covering the whole body, regulated to the temperature of 38 °C for 30 minutes.
  Interventions: Device: prewarming 30 minutes
- Standard care (No Intervention): warming with cotton sheet and blanket for 20 minutes.

INTERVENTIONS:
Device: prewarming 20 minutes — prewarming with a forced air warming system, using a blanket covering the whole body, regulated to the temperature of 38 °C for 20 minutes.
  Arms: Prewarming 20 minutes
Device: prewarming 30 minutes — prewarming with a forced air warming system, using a blanket covering the whole body, regulated to the temperature of 38 °C for 30 minutes.
  Arms: Prewarming 30 minutes

SUMMARY:
The present proposal intends to determine the effect of prewarming on body temperature in the perioperative period of patients submitted to digestive system surgeries and to evaluate a perioperative "Zero-Heat-Flux Cutaneous" body temperature thermometer in comparison to the standard care (temporal thermometer in the preoperative and postoperative, and esophageal in the intraoperative period). This is a randomized clinical trial consisting of three groups, namely: preoperative warming of patients with blanket and cotton sheet (control); preoperative warming with forced air warming system for 20 minutes (Intervention 1), and participants submitted to preoperative warming with a forced air warming system for 30 minutes (Intervention 2).

DETAILED DESCRIPTION:
The present proposal intends to determine the effect of prewarming on body temperature in the perioperative period of patients submitted to digestive system surgeries and to evaluate a perioperative "Zero-Heat-Flux Cutaneous" body temperature thermometer in comparison to the standard care (temporal thermometer in the preoperative and postoperative, and esophageal in the intraoperative period). This is a randomized clinical trial consisting of three groups, namely: preoperative warming of patients with blanket and cotton sheet (control); preoperative warming with forced air warming system for 20 minutes (Intervention 1), and participants submitted to preoperative warming with a forced air warming system for 30 minutes (Intervention 2)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over at the time of data collection
* Patients submitted to elective oncological surgery of the digestive, curative or palliative system, with anesthesia duration of at least one hour

Exclusion Criteria:

* Subjects with body temperature equal to or greater than 38 ºC at the time of admission to the Surgical Center
* Patients submitted to video laparoscopic or minimally invasive surgeries

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with temperature below 36 degrees measured by "Zero-Heat-Flux Cutaneous" body temperature thermometer | Perioperative period
  Number of patients with temperature below 36 degrees measured by "Zero-Heat-Flux Cutaneous" body temperature thermometer in comparison to number of patients with temperature below 36 degrees measured by the standard care (temporal thermometer in the preoperative and postoperative, and esophageal in the intraoperative period).

CONTACTS AND LOCATIONS:
Locations (1):
- ICESP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No